CLINICAL TRIAL: NCT06051396
Title: Phenotyping of the Out-of-proportion Pulmonary Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mahmoud Badwy, Assistant Lecturer, Assiut University
Other Study IDs: Assiut 3131
Record Dates: First submitted 2023-09-18; First posted 2023-09-22 (Actual); Last update posted 2023-11-24 (Actual); Status verified 2023-11

CONDITIONS: 1- Haemodynamic Phenotyping of the Out - of - Proportion PH to Guide Different Therapeutic Lines

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Right sided heart catheterization — Hemodynamic evaluation was performed in the supine position. RHC was performed using the modified Seldinger technique with an 8F sheath inserted in the jugular, basilic or cephalic vein . The Swan-Ganz catheter was a 7F, two-lumen, fluid filled, and pressure-measuring tipped catheter (Corodyn TD; Braun Medical, Bethlehem, PA, USA). The zero-level reference was determined at midthoracic line.(9)

SUMMARY:
Pulmonary hypertension (PH) is a pathophysiological disorder that may involve multiple clinical conditions and may be associated with a variety of cardiovascular and respiratory diseases. The complexity of managing PH requires a multidisciplinary approach, with active involvement of patients with PH in partnership with clinicians.(1) All age groups are affected. Present estimates suggest a PH prevalence of 1% of the global population. Due to the presence of cardiac and pulmonary causes of PH, prevalence is higher in individuals aged 65 years. Globally, LHD is the leading cause of PH. Lung disease, especially chronic obstructive pulmonary disease (COPD), is the second most common cause. In the UK, the observed PH prevalence has doubled in the last 10 years and is currently 125 cases/million inhabitants. (2) Pulmonary hypertension is defined by a mean pulmonary arterial pressure (mPAP) more than 20 mmHg at rest according to the 2022 ESC/ERS Guidelines for the diagnosis and treatment of pulmonary hypertension . It is essential to include PVR and pulmonary arterial wedge pressure (PAWP) in the definition of pre-capillary PH, in order to discriminate elevated PAP due to pulmonary vascular disease (PVD) from that due to left heart disease (LHD), elevated pulmonary blood flow, or increased intrathoracic pressure.(3) Clinical classification of pulmonary hypertension includes GROUP 1 Pulmonary arterial hypertension (PAH), GROUP 2 PH associated with left heart disease, GROUP 3 PH associated with lung diseases and/or hypoxia, GROUP 4 PH associated with pulmonary artery obstructions and GROUP 5 PH with unclear and/or multifactorial mechanisms. (3) Pulmonary hypertension is frequently observed in patients with COPD and/or emphysema, diffuse parenchymal lung diseases and hypoventilation syndromes. Pulmonary hypertension is uncommon in obstructive sleep apnoea unless other conditions coexist, such as COPD or daytime hypoventilation.

In patients with lung disease, PH is categorized as non-severe or severe, Whereas non-severe PH is common in advanced COPD and ILD defined by spirometric criteria, severe PH is uncommon, occurring in 1-5% of cases of COPD and ,10% of patients with advanced ILD, with limited data in obesity hypoventilation syndrome.(4) Pulmonary hypertension presenting in patients with lung disease may be due to a number of causes, including undiagnosed CTEPH or PAH. A number of distinct phenotypes of PH in patients with lung disease, including a pulmonary vascular phenotype, have been proposed. The pulmonary vascular phenotype is characterized by better preserved spirometry, low DLCO, hypoxaemia, a range of parenchymal involvement on lung imaging, and a circulatory limitation to exercise.(5) Cardiac comorbidities are also common in patients with lung disease and may contribute to increased risk for hospitalization, longer length of stay, pulmonary hypertension and CVD-related mortality.(6) A vast category of patients suffering from parenchymal lung diseases (often accompanied by minor pulmonary impairment on pulmonary function test and/or CT scan) with an unexplained severe degree of PH was brought to the attention of physicians. In these patients, the development of moderate to severe PH, which is disproportionate to the degree of parenchymal lung disease and hypoxia, has been termed "out-of-proportion" PH, and an arbitrary value of . 35 mm Hg mean pulmonary artery pressure has been selected to identify this category of patients.(7) and there is limited data about the Out-of proportion PH and it different phenotypes

ELIGIBILITY:
Inclusion Criteria:

* All Patients presented with severe pulmonary hypertension (PASP > 70mmHg by echocardiographic assessment) (8) associated with chronic lung diseas will be included in the study

Exclusion Criteria:

* 1- Age under 18 years. 2- Severe PH proportional to the disease. 3- Hemodynamically unstable condition requiring inotropic or vasoactive drugs. 4- Severe chest wall deformity. 5- Pregnant women. 6- Right-sided endocarditis, right-sided tumor, or thrombus. 7- Severe coagulopathy or bleeding diathesis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All Patients presented with severe pulmonary hypertension (PASP > 70mmHg by echocardiographic assessment) (8) associated with chronic lung diseas will be included in the study
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
1- Haemodynamic phenotyping of the out - of - proportion PH to guide different therapeutic lines | 2 yrs
  Identification of different phenotypes of severe pulmnary hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Badwy, specialist, Principal Investigator — Assiut University
Locations (1):
- Mahmoud Badwy, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Humbert M, Germany MMH, Berger RMF, Denmark JC, Germany EM, Germany BN, et al. 2022 ESC / ERS Guidelines for the diagnosis and treatment of pulmonary hypertension Developed by the task force for the diagnosis and treatment of ( ESC ) and the European Respiratory Society ( ERS ). Endorsed by the International Society for Heart and Lu. Eur Heart J. 2022;1-114.